CLINICAL TRIAL: NCT05531162
Title: Repetitive Gravitationnal Changes on the Body-environment Relationship
Brief Title: Body-environment Relationship Related Modified Gravity
Acronym: ENACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A01317-36
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Body Schema
Keywords: adaptation; cognition; extreme environment; confined environment; stress; performances; olfaction; somesthesia; space mission
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Intervention Model Description: a group of parabolic flyers with and without prior experience of microgravity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Microgravity condition (Other): a group of parabolic flyers exposed to micro and partial gravity
  Interventions: Other: Cognition and emotional neuropsychologicl evaluations

INTERVENTIONS:
Other: Cognition and emotional neuropsychologicl evaluations — Cognitive ans sensory performances during repetitive micro and partial gravity exposure

SUMMARY:
The overall objective of this study is to better understand the relationship between the body and its environment, including cognitive performance, following repeated changes in gravity, including microgravity (0G) and modified gravity (i.e., hypergravity (1.8G) and modified gravity (Martian gravity)

DETAILED DESCRIPTION:
On the eve of the next long voyages into space and the event of space tourism, it becomes more and more urgent to understand how to preserve the health of spacemen (i.e., by profession or by leisure). Extreme and unusual environments, and isolated and confined environments (EUE/ICE) are characterized by unique sensory stimulation. They are known to have negative effects on human psychology, cognitive abilities and physiology, threatening the outcome of space missions or travel. In addition, with the construction of the future Gateway base, the upcoming colonies to Mars and space tourism, travel from one point to another will be much more frequent. These raise new questions that will have to be addressed, whether it is the prolonged duration of a stay in a microgravity environment (i.e., absence of gravitational force between man and his support), in partial gravity and thus the issue of recovery from one trip to the next. These modifications of the environment imply the implementation of several adaptation processes to preserve the homeostatic capacity of the organism. This allows the organism to maintain a relatively stable internal state that persists despite external changes. Nevertheless, many questions remain unanswered. One such question is the impact of repeated changes in gravity during flight to the point of attachment (e.g., colony). The objective of the study is therefore to better understand the relationship between the body and its environment due to repeated changes in gravity, including microgravity.

Beyond that, these results will contribute to enrich the knowledge of this real human challenge that is the question of the adaptation of the human being to the constraints of space travel.

ELIGIBILITY:
Inclusion Criteria:

* Existence of an informed and written consent from the subject
* Not pregnant
* No anxiety disorder and/or depression
* Not to have suffered a head injury
* Have obtained a medical certificate of aptitude for parabolic flights
* Be affiliated to the French Social Security, or have a European Health Insurance Card or equivalent

Exclusion Criteria:

* Pregnant women, parturients and nursing mothers
* Endocrine pathology (e.g., hyperthyroidism, diabetes)
* High blood pressure
* History of head trauma, mood or cardiovascular disorders, cognitive impairment
* Recent illicit drug use
* Alcohol dependence
* Neurological disease and/or history of neurological disease Psychiatric disease and/or history of psychiatric disease
* Anti-inflammatory treatment
* Psychotropic treatment
* Treatments that interfere with heart rate (e.g., beta-blockers, calcium channel blockers, a1 receptor agonists)
* Persons deprived of liberty, persons hospitalized without consent, persons admitted to a health or social institution for purposes other than research (L-1121-5 to L-1121-8-1)
* Protected adults, adults unable to express their consent and not subject to a protective measure
* Participation in other simultaneous trials if this or these protocols concern a pharmacological clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-23 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Psychological data | one hour before the flight
  Freiburg Mindfulness Inventory questionnaire of 14 items (each item has a score from 1 to 4 i.e. minimal value 14 and maximal value 56, with a couple of reversed item to score)
Psychological data | one hour after the flight
  Freiburg Mindfulness Inventory questionnaire of 14 items (each item has a score from 1 to 4 i.e. minimal value 14 and maximal value 56, with a couple of reversed item to score)
stress | one hour before the flight
  Perceived Stress Scale questionnaire: 10 item-questionnaire to perceive stress (each item from 0 to 4: minimal value 0/no stress and maximal value 40 highest stress level)
stress | one hour after the flight
  Perceived Stress Scale questionnaire: 10 item-questionnaire to perceive stress (each item from 0 to 4: minimal value 0/no stress and maximal value 40 highest stress level)
Cognition | one hour before the flight
  Cognitive test battery questionnaire, 2D and 3D testing during one session: three scores ponderated (each with 6 plots represented with a spider graph measuring the surface from arbitrary unit)
Cognition | one hour after the flight
  Cognitive test battery questionnaire, 2D and 3D testing during one session: three scores ponderated (each with 6 plots represented with a spider graph measuring the surface from arbitrary unit)
Olfaction | one hour before the flight
  Olfactive discrimination test
Olfaction | one hour after the flight
  Olfactive discrimination test
Posture | one hour before the flight
  Ellipse of the center of gravity measurment
Posture | one hour after the flight
  Ellipse of the center of gravity measurment
Physiological data | Continuous recording all along microgravity exposure up to 1hour after the end of the flight
  Heart Rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No